CLINICAL TRIAL: NCT02589821
Title: A Randomized, Double-blind, Multi-center Phase III Clinical Study to Assess the Efficacy and Safety of Surufatinib Compared to Placebo in Patients With Advanced Pancreatic Neuroendocrine Tumors
Brief Title: Phase III Study of Surufatinib in Treating Advanced Pancreatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-012-00CH3
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — surufatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surufatinib (Experimental): Surufatinib 300 mg, orally, once daily (QD)
  Interventions: Drug: Surufatinib
- Placebo (Placebo Comparator): Placebo 300 mg, orally, once daily (QD)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Surufatinib — Surufatinib 300 mg once a day (QD) will be orally administrated on a 28-day cycle
  Other Names: HMPL-012; Sulfatinb
  Arms: Surufatinib
Other: Placebo — Placebo 300 mg once a day (QD) will be orally administrated on a 28-day cycle
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo controlled, multi-center Phase III study to assess the efficacy of Surufatinib 300 mg once a day in treating advanced pancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
195 patients will be randomly assigned (in 2:1 ratio) to the Surufatinib or Placebo treatment group based on interactive web response system（IWRS).The patients will receive continuous oral treatment, every 28-day treatment cycle until progression of disease occurs, intolerable toxicity or other protocol specified end-o-treatment criteria is met. The tumor should be assessed every 8 weeks (+/-3 days) within the first year and every 12 weeks (+/-3 days) after the patient has been treated for one year.

A Blinded Independent Image Review Committee (BIIRC) will subsequently provide a central review of the oncologic imaging materials from the patients.

An independent Data Monitoring Committee (IDMC) will be assembled to monitor safety and efficacy data, and evaluate interim analysis. If the interim analysis demonstrates overwhelming efficacy of the treatment arm with respect to PFS (primary endpoint) versus control arm, IDMC could recommend terminating and to unblinding the study and sulfatinib will be offered to the control arm patients who are still on treatment until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Adequately understand the study and voluntarily sign the Informed Consent Form;
2. Be at least 18 years old;
3. Based on central pathology review results, patients have a confirmed histologically pathology diagnosis of low- or intermediate grade (G1 or G2) advanced (unresectable or distant metastatic) PNET. G1 is defined as < 2 mitoses /10 high-power field［HPF］and/or <3% Ki-67 index; G2 is defined as 2-20/10 HPF and/or 3-20% Ki-67 index. If the mitotic ratio and Ki-67 index correspond to different grade, the higher grade should be used to assign classification.
4. Have previously progressed on no more than two types of systemic anti-tumor therapy, including long-acting somatostatin analogs (SSAs), interferon, PRRT(peptide receptor radionuclide therapy), mTOR inhibitors or chemotherapy(chemotherapies were considered as one kind of regimen, regardless of medications and cycles); patients who are unable or unwilling to receive such treatments are also eligible;
5. Patients must have radiological documentation of progression of disease within 12 months prior to randomization.
6. Have measurable lesions (according to RECIST 1.1);
7. Absolute neutrophil count (ANC) of ≥1.5×109/L, platelet count of ≥100×109/L, and hemoglobin ≥9 g/dL;
8. Serum total bilirubin <1.5 times the upper limit of normal (ULN);
9. Patients who do not have liver metastasis, with alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤ 2.5 times the ULN; and who do have liver metastatic, with ALT and AST ≤ 5 times ULN.
10. Serum creatinine <1.5 times ULN and creatinine clearance ≥60 ml/min;
11. International Normalized Ratio (INR) ≤1.5 ULN and activated partial thromboplastin time (APTT) ≤1.5 ULN.
12. Have a performance status (PS) of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale;
13. Have expected survival of more than 12 weeks;
14. Male or females patients with reproductive potential must agree to use an effective contraceptive method, for example, double-barrier device, condom, oral or injected birth control medication or intrauterine device, during the study and within 90 days after study treatment discontinuation. All female patients are considered to be fertile, unless the patient had natural menopause or artificial menopause or sterilization (such as hysterectomy, bilateral oophorectomy or ovarian irradiation).

Exclusion Criteria:

1. High grade (G3) neuroendocrine cancer, adenocarcinoid, pancreatic islet cell carcinoma, goblet cell carcinoid, large cell neuroendocrine carcinoma and small cell carcinoma;
2. Functional NETs which need to be treated with long acting SSAs to control disease related syndromes, such as insulinoma, gastrinoma, glucagonoma, somatostatinoma, ACTHoma, VIPoma, accompanied by carcinoid syndrome, Zollinger-Ellison syndrome or other active symptoms;
3. Have received anti-VEGF/VEGFR targeted drugs and progressed upon these drugs;
4. Urinalysis shows urine protein ≥ 2+ or 24-hour protein quantity test shows urinary protein ≥1 g;
5. Serum potassium, calcium (albumin-bound ionic or corrected) or magnesium exceeds the normal range with clinical significance;
6. Under anti-hypertension treatment, still uncontrolled hypertension, defined as: systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg;
7. Gastrointestinal disease or condition that investigators suspect may affect drug absorption, including, but not limited to, active gastric and duodenal ulcers, ulcerative colitis and other digestive disease, gastrointestinal tumor with active bleeding, or other gastrointestinal conditions that may cause bleeding or perforation by investigator's discretion;
8. History or presence of a serious hemorrhage (>30 ml within 3 months), hemoptysis (>5 ml blood within 4 weeks) or a thromboembolic event (including transient ischemic attack) within 12 months;
9. Clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction within 6 months prior to enrollment, severe/unstable angina pectoris or coronary artery bypass grafting, congestive heart failure according to the New York Heart Association (NYHA) classification ≥ 2; ventricular arrhythmias which needs drug treatment; LVEF (LVEF) <50%;
10. Mean corrected QT interval (QTc) ≥ 480 msec;
11. Other malignancies diagnosed within the previous 5 years, except basal cell carcinoma or cervical carcinoma in situ after radical resection;
12. Anti-tumor therapy received within 4 weeks prior to the initiation of the investigational treatment, including, but not limited to, chemotherapy, radical radiotherapy, targeted therapy, immunotherapy and anti-tumor Chinese medicine treatment, hepatic chemoembolization, cryoablation and radiofrequency ablation ;
13. Palliative radiotherapy for a bone metastasis lesion within 2 weeks prior to the initiation of the investigational treatment;
14. Drugs containing St John's wort taken within 3 weeks prior to the first study treatment, or other strong inducers with CYP3A4 or strong inhibitors taken within two weeks prior to the first study treatment (see appendix 3);
15. Any clinically significant active infection, including, but not limited to, human immunodeficiency virus (HIV) infection;
16. History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×104/ml); known Hepatitis C virus infection with HCV RNA positive (copies ≥1×103/m); or liver cirrhosis, etc.
17. Surgery (except biopsy) within 28 days prior to the initiation of investigational treatment or unhealed surgical incision; 18 Brain metastases and/or spinal cord compression not treated by surgery and/or radiotherapy, and with no clinical imaging evidence of disease stability;

19. Toxicity from a previous anti-tumor treatment that does not return to Grade 0 or 1 (except for hair loss); 20. Received investigational treatments in other clinical studies within 4 weeks prior to enrollment; 21. Women who are pregnant or lactating; 22. Other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions are inappropriate for the use of the investigational product or affect interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2015-12-07 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 7 months after the last patient enrolled
  the duration between the randomization date and the first disease progression (PD) or death (whichever comes first).

SECONDARY OUTCOMES:
The objective response rate of the tumor (ORR) | 7 months after the last patient enrolled
  the incidence of confirmed complete response or partial response
The disease control rate (DCR) | 7 months after the last patient enrolled
  the incidence of complete response, partial response and stable disease
Duration of Response (DoR) | 7 months after the last patient enrolled
  the duration between the date the criteria for complete response or partial response was first measured (first record shall prevail) and the date of disease recurrence or progression as objectively recorded
Time to Response (TTR) | 7 months after the last patient enrolled
  the period from the date of randomization to the date when the criteria for complete response or partial response was first measured (first record shall prevail).
Overall survival (OS) | 7 months after the last patient enrolled
  the time from the date of randomization to the date of death (all causes)
•adverse events evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 | From first dose to within 30 days after the last dose
  The safety and tolerability of Surufatinib will be evaluated based on adverse events data. Other safety parameters include physical examination, vital signs, laboratory test results (i.e., hematology, chemistry panel, and urinalysis), 12-lead electrocardiogram, and ultrasonic cardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Songhua Fan, MD, Study Director — Hutchison Medi Pharma
Locations (5):
- China (5):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - the 307 Hospital of People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - West China Hospital, Sichuan University, Chengdu, Sichuan

REFERENCES:
- [Derived] Xu J, Shen L, Li J, Zhou Z, Bai C, Li Z, Chi Y, Li E, Yu X, Xu N, Bai Y, Wang X, Yuan X, Liu T, Yin Y, Chen J, Hu H, Li X, Xiu D, Zhang T, Lou W, Ying J, Qin S, Deng Y, Tao M, Cheng Y, Fan S, Luo X, Guo X, Shi MM, Su W. Surufatinib in advanced neuroendocrine tumours: Final overall survival from two randomised, double-blind, placebo-controlled phase 3 studies (SANET-ep and SANET-p). Eur J Cancer. 2025 Jun 3;222:115398. doi: 10.1016/j.ejca.2025.115398. Epub 2025 Mar 30. PMID 40306120
- [Derived] Li J, Cheng Y, Bai C, Xu J, Shen L, Li J, Zhou Z, Li Z, Chi Y, Yu X, Li E, Xu N, Liu T, Lou W, Bai Y, Yuan X, Wang X, Yuan Y, Chen J, Guan S, Fan S, Su W. Health-related quality of life in patients with advanced well-differentiated pancreatic and extrapancreatic neuroendocrine tumors treated with surufatinib versus placebo: Results from two randomized, double-blind, phase III trials (SANET-p and SANET-ep). Eur J Cancer. 2022 Jul;169:1-9. doi: 10.1016/j.ejca.2022.03.027. Epub 2022 Apr 28. PMID 35489301
- [Derived] Li J, Cheng Y, Bai C, Xu J, Shen L, Li J, Zhou Z, Li Z, Chi Y, Yu X, Li E, Xu N, Liu T, Lou W, Bai Y, Yuan X, Wang X, Yuan Y, Chen J, Guan S, Fan S, Su W. Treatment-related adverse events as predictive biomarkers of efficacy in patients with advanced neuroendocrine tumors treated with surufatinib: results from two phase III studies. ESMO Open. 2022 Apr;7(2):100453. doi: 10.1016/j.esmoop.2022.100453. Epub 2022 Mar 25. PMID 35344750
- [Derived] Xu J, Shen L, Bai C, Wang W, Li J, Yu X, Li Z, Li E, Yuan X, Chi Y, Yin Y, Lou W, Xu N, Bai Y, Zhang T, Xiu D, Wang X, Yuan Y, Chen J, Qin S, Jia R, Lu M, Cheng Y, Zhou Z, Li J, He J, Su W. Surufatinib in advanced pancreatic neuroendocrine tumours (SANET-p): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Nov;21(11):1489-1499. doi: 10.1016/S1470-2045(20)30493-9. Epub 2020 Sep 20. PMID 32966810